CLINICAL TRIAL: NCT04383223
Title: iTransition: Pilot Testing a Multilevel Technology Based Intervention to Support Youth Living With HIV From Adolescent to Adult Care
Brief Title: iTransition Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Sophia Hussen, Assistant Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00114532; R34MH116805-01A1 (NIH)
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Results first posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Human Immunodeficiency Virus; HIV Seropositivity
Keywords: HIV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Seropositivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- YLH Historical Control Group (No Intervention): Participants in this group will have the following phases:
  * Screening
  * Single visit assessment
- YLH iTransition Intervention Group (Experimental): Participants in this group will have the following phases:
  * Screening
  * Baseline Visit
  * Follow-Up visits at 6, 12 and 18 month
  * Interview visits for selected YLH around 3 and 9 month
  Interventions: Behavioral: iTransition
- Provider Group (Experimental): Participants in this group will have the following phases:
  * Screening
  * Baseline Visit
  * Follow-Up visits at 6, 12 and 18 month
  * Interview visits for selected YLH around 3, 9 and 15 month
  Interventions: Behavioral: iTransition
- Transition Champion Group (Experimental): Participants in this group will have the following phases:
  * Screening
  * Baseline Visit and Follow-Up visits at 6, 12 and 18 month
  * Interview visits for selected YLH around 3, 9 and 15 month
  Interventions: Behavioral: iTransition

INTERVENTIONS:
Behavioral: iTransition — Is a mobile website application (app), and it can be used on a range of devices (computer, tablet, smartphone) and operating systems (iOS, Android, Windows). Features of iTransition will include, but are not limited to: medication reminders, calendar tracking of appointments, direct messaging between youth and providers, and privacy password lock.
  Arms: Provider Group; Transition Champion Group; YLH iTransition Intervention Group

SUMMARY:
Youth living with HIV are at high risk of falling out of care when they transition from pediatric to adult care. The investigators are proposing to develop a mobile app to help both clinical providers and patients navigate this process.

DETAILED DESCRIPTION:
The transition from pediatric/adolescent to adult-oriented care settings can be disruptive to care engagement for youth living with HIV (YLH).

The objective of this trial is to pilot and evaluate effectiveness of iTransition, an mHealth intervention to improve healthcare transition (HCT) at the patient, provider, and clinic levels.It is a prospective non-randomized intervention pilot trial of subjects in Atlanta, GA and Philadelphia, PA: around 100 YLH (50 intervention and 50 historical controls), 20 providers, and 8 Transition Champions. The study duration is 12 and 18 months for YLH and provider/champions, respectively.

At baseline, YLH ≥18 years planning for care transition within 6 months, and reporting consistent internet access. Providers and Transition Champions must report working with transitioning YLH at pediatric/adolescent and/or adult HIV care centers.

Data measures include iTransition usage, intervention satisfaction and health surveys, interviews (select participants), and medical chart review to measure clinical outcomes. The primary clinical outcome variable, measured at the patient-level (YLH), is linkage to adult care (defined dichotomously as having one completed adult clinic appointment or not). Secondary clinical outcomes are care retention (dichotomously defined as having or not having one visit in each 6-month period) and viral suppression (<200 copies/ml) at 1-year post-baseline visit.

ELIGIBILITY:
Inclusion Criteria:

For YLH Historical Control Group

* YLH (regardless of gender/assigned sex at birth) age ≥ 18 years;
* Has plan for HCT within next 6 months;
* Enrolled in care at Grady IDP pediatric/adolescent clinic or CHOP AI/SI clinics.

For YLH iTransition Intervention Group

* YLH (regardless of gender/assigned sex at birth) age ≥ 18 years;
* Has plan for HCT within next 6 months;
* Enrolled in care at Grady IDP pediatric/adolescent clinic or CHOP AI/SI clinics;
* Owns a smartphone and/or tablet
* Reports consistent internet access (defined as no lapse >24 hours in last 6 months) via their smartphone or tablet.

For Provider Group

* Staff member at Grady IDP (pediatric/adolescent clinic, adult women's clinic, and/or adult men's clinic), CHOP AI/SI clinics, UPHS: HUP or Presby infectious disease clinics;
* Works with transitioning YLH;
* Access to internet via any device (e.g., smartphone, tablet, computer);
* Endorse participation in the HCT process.

For Transition Champion Group

* Staff member at Grady IDP (pediatric/adolescent clinic, adult women's clinic, and/or adult men's clinic), CHOP AI/SI clinics, UPHS: HUP or Presby infectious disease clinics;
* Works with transitioning YLH;
* Endorse participation in the HCT process;
* Access to internet via any device (e.g., smartphone, tablet, computer);
* Nominated by clinic staff where employed to be iTransition intervention point person (champion).

Exclusion Criteria For YLH Historical Control Group

* Youth who are <18 years old;
* Youth who are not living with HIV;
* Transition is not expected (from pediatric/adolescent to adult care) within the next 6 months;
* Presence of serious psychiatric symptoms (e.g., active hallucinations, thought disorder) that would impair the individual's ability to provide true informed consent or participate in the study activities;
* Visibly distraught (e.g., suicidal, homicidal, exhibiting violent behavior) at the time of consent.

For YLH iTransition Intervention Group

* Youth who are <18 years old;
* Youth who are not living with HIV;
* Transition is not expected (from pediatric to adult care) within the next 6 months;
* Does not own smartphone/tablet and has inconsistent internet access (i.e. has had one or more lapse >24 hrs in the last three months);
* Presence of serious psychiatric symptoms (e.g., active hallucinations, thought disorder) that would impair the individual's ability to provide true informed consent or participate in the study activities;
* Visibly distraught (e.g., suicidal, homicidal, exhibiting violent behavior) at the time of consent.

For Provider Group

* Not a staff member at Grady IDP, CHOP SI/AI, UPHS: HUP or Presby infectious disease clinics;
* Does not work with transitioning YLH;
* Does not have access to internet via any device (e.g., smartphone, tablet, computer).

For Transition Champion Group

* Not a staff member at Grady IDP, CHOP SI/AI, UPHS: HUP or Presby infectious disease clinics;
* Does not work with transitioning YLH;
* Does not have access to internet via any device (e.g., smartphone, tablet, computer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Hussen, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Grady Hospital, Atlanta, Georgia
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania Health System - HUP and Presby infectious disease clinics, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Survey data will be shared as well as de-identified clinical outcome data Study protocols and statistical analysis plans upon request
Supporting Information: Study Protocol, SAP
Time Frame: Data is expected to become available in September 2022 upon completion of the study.
Access Criteria: Data will not be deposited into a public repository, but will be made available upon request to the principal investigator. The PI will discuss requests with the other study team members, and make a determination about whether data can be shared.

RESULTS

PARTICIPANT FLOW:
Groups:
- YLH iTransition Intervention Group: Participants in this group will have the following phases:
  * Screening
  * Baseline Visit
  * Follow-Up visits at 6, 12 and 18 month
  * Interview visits for selected YLH around 3 and 9 month
  iTransition: Is a mobile website application (app), and it can be used on a range of devices (computer, tablet, smartphone) and operating systems (iOS, Android, Windows). Features of iTransition will include, but are not limited to: medication reminders, calendar tracking of appointments, direct messaging between youth and providers, and privacy password lock.
- Provider Group: Participants in this group will have the following phases:
  * Screening
  * Baseline Visit
  * Follow-Up visits at 6, 12 and 18 month
  * Interview visits for selected YLH around 3, 9 and 15 month
  iTransition: Is a mobile website application (app), and it can be used on a range of devices (computer, tablet, smartphone) and operating systems (iOS, Android, Windows). Features of iTransition will include, but are not limited to: medication reminders, calendar tracking of appointments, direct messaging between youth and providers, and privacy password lock.
- Transition Champion Group: Participants in this group will have the following phases:
  * Screening
  * Baseline Visit and Follow-Up visits at 6, 12 and 18 month
  * Interview visits for selected YLH around 3, 9 and 15 month
  iTransition: Is a mobile website application (app), and it can be used on a range of devices (computer, tablet, smartphone) and operating systems (iOS, Android, Windows). Features of iTransition will include, but are not limited to: medication reminders, calendar tracking of appointments, direct messaging between youth and providers, and privacy password lock.
Period: Overall Study
Arm/Group | YLH Historical Control Group | YLH iTransition Intervention Group | Provider Group | Transition Champion Group
Started | 21 | 33 | 17 | 7
Completed | 21 | 33 | 17 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | YLH Historical Control Group | YLH iTransition Intervention Group | Provider Group | Transition Champion Group | Total
Number analyzed (Participants) | 21 | 33 | 17 | 7 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.73 (0.94) | 24.64 (1.03) | 41.47 (7.71) | 39.00 (6.00) | 29.62 (0.97)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 7 | 3 | 12 | 4 | 26
  Male | 13 | 28 | 5 | 3 | 49
  Non-binary | 1 | 2 | 0 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 0 | 3
  Not Hispanic or Latino | 20 | 33 | 15 | 7 | 75
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 16 | 31 | 5 | 2 | 54
  White | 1 | 1 | 8 | 4 | 14
  More than one race | 4 | 0 | 0 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 21 | 33 | 17 | 7 | 78

OUTCOME MEASURES:

1. Primary Outcome: Linkage to Adult Care
Description: Defined dichotomously as having one completed adult clinic appointment or not.
Time Frame: 18 month post-intervention
Population: This outcome only applies to the groups with YLH (Youth Living With HIV) participants.
Measure: Count of Participants; unit: Participants
Arm/Group | YLH Historical Control Group | YLH iTransition Intervention Group | Provider Group | Transition Champion Group
Number analyzed (Participants) | 21 | 33 | 0 | 0
Participants | 16 | 22 | 0 | 0

2. Secondary Outcome: Care Retention Per Each 6-month Period
Description: Defined dichotomously as having one completed medical visit in each 6-month period.
Time Frame: Baseline, 6 month post-intervention, 12 month post-intervention, 18-month post-intervention
Population: This outcome only applies to the groups with YLH (Youth Living With HIV) participants.
Measure: Count of Participants; unit: Participants
Arm/Group | YLH Historical Control Group | YLH iTransition Intervention Group | Provider Group | Transition Champion Group
Number analyzed (Participants) | 21 | 33 | 0 | 0
Participants
  Number of participants with one completed medical visit from Baseline to 6 month post-intervention | 17 | 27 | 0 | 0
  Number of participants with one completed medical visit from 6 to 12 month post-intervention | 14 | 31 | 0 | 0
  Number of participants with one completed medical visit from 12 to 18 month post-intervention | 16 | 22 | 0 | 0

3. Secondary Outcome: Number of Participants With Viral Suppression
Description: Viral suppression is defined as <200 copies/ml blood at 1-year post-baseline.
Time Frame: Baseline, 1-year post-intervention
Population: This outcome only applies to the groups with YLH (Youth Living With HIV) participants.
Measure: Count of Participants; unit: Participants
Arm/Group | YLH Historical Control Group | YLH iTransition Intervention Group | Provider Group | Transition Champion Group
Number analyzed (Participants) | 21 | 33 | 0 | 0
Participants | 10 | 26 | 0 | 0

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the time of the intervention and continuing through the end of the study, at 18 months post-intervention.
Arm/Group | YLH Historical Control Group | YLH iTransition Intervention Group | Provider Group | Transition Champion Group
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/33 | 0/17 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/33 | 0/17 | 0/7
Other Adverse Events (participants affected / at risk) | 0/21 | 0/33 | 0/17 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-08-11): https://cdn.clinicaltrials.gov/large-docs/23/NCT04383223/Prot_001.pdf
  • Informed Consent Form (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/23/NCT04383223/ICF_000.pdf